CLINICAL TRIAL: NCT00147342
Title: The Effect of Basal Insulin During Exercise on the Development of Hypoglycemia in Children With Type 1 Diabetes
Brief Title: The Effect of Insulin During Exercise on the Development of Low Blood Sugar in Individuals With Type I Diabetes
Status: Completed | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: DirecNet 007; HD041890; HD041906; HD041918; HD041915; HD041908; HD041919
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type I
Keywords: exercise; hypoglycemia; Diabetes Mellitus, Type I; glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Most children with type 1 diabetes have a drop in the blood sugar during exercise. This drop in the blood sugar can result in hypoglycemia (low blood sugar). In children using an insulin pump, there is an opportunity to reduce the basal insulin rate during exercise. This study is being conducted to determine if decreasing the insulin that is received during exercise will reduce the risk of hypoglycemia. We hope to learn more about how the body responds to hypoglycemia and to hyperglycemia (high blood sugar) when it occurs.

As part of the study, children will have a visit on two different days. During each visit, children will exercise on a treadmill for about 60 minutes. During one of the visits, the children's basal rate will be continued during the exercise. During one visit, the basal insulin will be stopped. The blood sugar will be checked frequently during the exercise.

DETAILED DESCRIPTION:
Each child will have two study visits. The visits will be between 1 and 4 weeks apart. The child will come to the research unit at the hospital at about 11:30 a.m. and will have lunch in the clinic.

* If the child has had a severe hypoglycemia episode in the 2 weeks before a visit or is ill at the time of either visit, the visit will be rescheduled.

The parent and child will be asked if they want to use a meter to test the child's hemoglobin A1c at home. If they want to do this, they will be given the meter and asked to test the child's A1c two times on the day before one of the visits. The two tests will be done at the same time and they will also be asked to check the child's blood sugar at the same time. The test involves a fingerstick similar to testing the blood sugar level with a home glucose meter.

At the start of each visit, a continuous glucose sensor will be inserted under the skin. This is done either in the stomach area, side, or buttock depending on which area looks like it will work best for the child. A special cream may be used to numb the skin before this sensor is placed. At the end of each visit, the child will have the option of removing the sensor or wearing it home for continued use.

During each visit, blood samples will be drawn frequently to measure glucose and other hormones. To make the blood sampling easier, a small tube, called a catheter, will be placed in a vein in the child's arm. A special cream may be used to numb the skin before the tube is placed. The tube will stay in the vein while the child is in the hospital. There may be some itching, stinging or pain from having the tube in the vein. However, there should be no pain when blood is drawn through the tube. If the tube stops working, a new one will need to be inserted.

* Blood sugar measurements will also be made with a home glucose meter. Instead of doing fingersticks, blood may be taken from the tube to measure the blood glucose with the home glucose meter.
* Blood samples will be taken and sent to a lab before, during, and after the exercise.
* In all, there will be 24 blood samples taken (12 samples during each of the visits).

During each visit, the child will be asked to walk on a treadmill.

* Before and after walking on the treadmill, the child will be checked for urine and blood ketones.
* During each visit, in the late afternoon, the child will walk on the treadmill for 15 minutes followed by a 5-minute rest period. This cycle of 15 minutes of exercise followed by a 5-minute rest period will be repeated 3 times for a total of 75 minutes.
* During one of the visits, the child's basal insulin rate will be stopped at the start of the exercise session and will be restarted about 45 minutes after the child stops exercising. During the other visit, the basal rate will be continued. A process like flipping a coin is used to decide the order of the visits.
* For both visits, the blood sugar needs to be between 120 and 200 at the start of the exercise. Between lunch and 4 p.m., the blood sugar will be checked a few times. To lower the blood sugar to this range, the child may be given insulin through the catheter to be used to draw the blood samples. No bolus insulin doses will be given with the child's pump after lunch. If the study doctors or nurses think the child's blood sugar may be too low to start exercise, a snack may be given to get the blood sugar to be in this range. If the blood sugar is too high or too low and cannot be corrected quickly enough, the exercise for that day may be postponed. If this happens, the child will need to return on another day.
* About 30 minutes after the exercise has ended, the child's blood sugar will be checked. If it is less than 250 mg/dL, a snack will be given and the last blood draw for the study will be made 15 minutes later. If the blood sugar is 250 mg/dL or higher, no snack will be given and the child's blood sugar will be checked in 15 minutes. At that time the child's insulin pump will be started if it was stopped, and a correction dose of insulin may be given.
* If at anytime after the exercise session the child's blood sugar is 325 mg/dL or higher, the child's insulin pump will be started and a correction dose of insulin may be given.

During each visit, the child's blood sugar will be checked frequently. If the blood sugar drops to 65 mg/dL or lower, the hypoglycemia will be treated with carbohydrate. The child will not be treated if the blood sugar is higher than 65 mg/dL.

Dinner will be given to the child at about 6:00 p.m. A bedtime snack will be given to the child to take home. The snack will be based on what the child would normally eat on a day with exercise.

The child will be instructed to not have any more exercise for the rest of the day. The child will be given a home glucose meter and asked to check his or her blood sugar prior to the bedtime snack, at midnight, 3 a.m., and before breakfast the next morning. The child will be asked to treat any blood sugars 80 mg/dL or lower and to record the information on a log that will be provided.

If the parent and child decided to do the A1c meter study at home, at one of the visits the study staff will check the A1c using the meter and the DCA2000. A fingerstick blood sample will also be sent to the central laboratory. The child's blood sugar will also be checked at the time of the tests.

The catheter for the blood draws will be removed and each visit will end at about 6:30 p.m.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes for at least 18 months (The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.)
* HbA1c <10.0% (The DCA2000 will be used to assess eligibility.)
* Age 8.0 to <18.0 years
* Weight >39.5 kg at reinfusion centers and >46.0 kg at discard centers
* BMI >5th and <95th percentiles for age and gender
* Stable insulin regimen for at least 1 month and not anticipating a change prior to the subject's completion of the study (Stable is defined as no change in the overall insulin program, i.e., no change from SC injections to pump.)
* Insulin regimen involves use of an insulin pump
* Normal thyroid function (measured within the previous year)

Exclusion Criteria:

* A recent injury to body or limb, Addison's disease, muscular disorder, use of any medication or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the exercise protocol
* Asthma which has been medically treated within the last year
* Current use of glucocorticoid medication (by any route of administration)
* Current use of a beta blocker medication
* Use of pseudoephedrine 48 hours prior to visit (if used in the 48 hours prior to the scheduled visit, the visit will be deferred)
* Severe hypoglycemia resulting in seizure or loss of consciousness in the 2 weeks prior to a visit (if a severe episode occurs within 2 weeks prior to the scheduled visit, the visit will be deferred)
* Active infection (if at the time of the scheduled visit an infection is present, the visit will be deferred)
* Anticipating a significant change in exercise regimen between visits (i.e. starting or stopping an organized sport)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55
Dates: Start 2005-05; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: William V Tamborlane, M.D., Study Chair — Department of Pediatrics, Yale University School of Medicine
Locations (6):
- United States (6):
  - Division of Pediatric Endocrinology and Diabetes, Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, University of Colorado, Aurora, Colorado
  - Department of Pediatrics, Yale University School of Medicine, New Haven, Connecticut
  - Nemours Children's Clinic, Jacksonville, Florida
  - Jaeb Center for Health Research, Tampa, Florida
  - Department of Pediatrics, University of Iowa Carver College of Medicine, Iowa City, Iowa

REFERENCES:
- [Result] Diabetes Research in Children Network (DirecNet) Study Group; Tsalikian E, Kollman C, Tamborlane WB, Beck RW, Fiallo-Scharer R, Fox L, Janz KF, Ruedy KJ, Wilson D, Xing D, Weinzimer SA. Prevention of hypoglycemia during exercise in children with type 1 diabetes by suspending basal insulin. Diabetes Care. 2006 Oct;29(10):2200-4. doi: 10.2337/dc06-0495. PMID 17003293
- [Result] Fox L, Dontchev M, Ruedy K, Beck R, Kollman C, Messer L, Coffey J, Wilson D, Doyle E, Tamborlane W, Steffes M; DirecNet Study Group. Relative inaccuracy of the A1cNow in children with type 1 diabetes. Diabetes Care. 2007 Jan;30(1):135-7. doi: 10.2337/dc06-0972. No abstract available. PMID 17192346